CLINICAL TRIAL: NCT02294006
Title: Activity and Safety of Everolimus in Combination With Octreotide LAR and Metformin in Patients With Advanced Pancreatic Well-differentiated Neuroendocrine Tumors (pWDNETs): a Phase II, Open, Monocentric, Prospective Study
Brief Title: Activity and Safety of Everolimus+Octreotide LAR+Metformin in Advanced Pancreatic Well-differentiated NETs
Acronym: MetNET1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ist Nazionale Tumori Milano
Record Dates: First submitted 2014-10-29; First posted 2014-11-19 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Well Differentiated Pancreatic Endocrine Tumor
Keywords: pancreatic; neuroendocrine; everolimus; metformin; octreotide
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — Everolimus; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- everolimus+octreotide LAR+metformin (Experimental): everolimus+octreotide LAR+metformin
  Interventions: Drug: Everolimus plus Octreotide LAR plus Metformin

INTERVENTIONS:
Drug: Everolimus plus Octreotide LAR plus Metformin — Everolimus plus Octreotide LAR plus Metformin

SUMMARY:
Abnormal PI3K-Akt-mTOR (mammalian target of rapamycin) pathway signaling and autocrine activation of the mTOR pathway, mediated through insulin-like growth factor 1 (IGF1), has been implicated in the proliferation of pNET ( primitive neuroectodermal tumor) cells. Everolimus ,an mTOR inhibitor (a central regulator of growth/proliferation, cellular metabolism and angiogenesis) has shown antitumor benefit in pNETs alone and in combination with Octreotide LAR in RADIANT-1 and RADIANT-3 studies.

Despite EVE-based phase II/III trials improve progression-free survival (PFS) for pNETs, they are limited to significantly prolong overall survival (OS). Metformin has recently shown some anti-cancer activity, both in vitro and in vivo studies by antisecretory properties to decrease insulin and IGF1 levels; and by antitumor effect due to AMPK (adenosine monophosphate kinase) activation and consequently inhibition to TSC1(tuberous sclerosis complex 1) -2/mTOR complex, mediated to LKB1 oncogene expression. The investigators retrospective experience, despite in a limited group of pWDNET, highlights the role of MET to improve clinical benefit in diabetic pts receiving EVE-OCT (octreotide) combination.

This study will investigate the antiproliferative potential of MET in combination with EVE and OCT in pWDNETs. MetNET1 prospective trial (EudraCT 2014-000888-41) may be helpful to either confirm or discard these preliminary findings.

The main objective of this study is to evaluate progression free survival rate at 12 months of treatment. The secondary objectives are safety, overall survival, response rate evaluation.

A sub-study analysis will evaluate circulant biomarkers levels (IL 6, IGF1) in blood samples.

DETAILED DESCRIPTION:
Abnormal PI3K-Akt-mTOR (mammalian target of rapamycin) pathway signaling and autocrine activation of the mTOR pathway, mediated through insulin-like growth factor 1 (IGF1), has been implicated in the proliferation of pNET ( primitive neuroectodermal tumor) cells. Everolimus ,an mTOR inhibitor (a central regulator of growth/proliferation, cellular metabolism and angiogenesis) has shown antitumor benefit in pNETs alone and in combination with Octreotide LAR in RADIANT-1 and RADIANT-3 studies.

Despite EVE-based phase II/III trials improve progression-free survival (PFS) for pNETs, they are limited to significantly prolong overall survival (OS). Metformin has recently shown some anti-cancer activity, both in vitro and in vivo studies by antisecretory properties to decrease insulin and IGF1 levels; and by antitumor effect due to AMPK (adenosine monophosphate kinase) activation and consequently inhibition to TSC1(tuberous sclerosis complex 1) -2/mTOR complex, mediated to LKB1 oncogene expression. The investigators retrospective experience, despite in a limited group of pWDNET, highlights the role of MET to improve clinical benefit in diabetic pts receiving EVE-OCT (octreotide) combination.

This study will investigate the antiproliferative potential of MET in combination with EVE and OCT in pWDNETs. MetNET1 prospective trial (EudraCT 2014-000888-41) may be helpful to either confirm or discard these preliminary findings.

The main objective of this study is to evaluate progression free survival rate at 12 months of treatment. The secondary objectives are safety, overall survival, response rate evaluation.

A sub-study analysis will evaluate circulant biomarkers levels (IL 6, IGF1) in blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of written informed consent (approved by the Institutional Ethics Committee Independent ) obtained after a careful study of screening procedures
2. Age >= 18 years old.
3. Patients with histological evidence of pNET well-differentiated G1 -G2
4. Configurable tumor disease (according to RECIST (Response Evaluation Criteria In Solid Tumors) ) .
5. Karnofsky Performance Status >= 60%.
6. Life expectancy greater than 6 months.
7. Is permitted to enroll patients who have not received any treatment for advanced disease or patients pretreated with surgery , chemotherapy or somatostatin analogues .
8. Basal blood tests :

   * Counts of neutrophils in absolute value > 1.5 x 109 / L.
   * Platelet count > 100 x 109 / L.
   * Hemoglobin > 9 g / dl .
   * Total Bilirubin < 1.5 times the upper limit of normal .
   * AST( aspartate aminotransferase), ALT (alanine aminotransferase)<2.5 times the upper limit of normal in patients without evidence of liver metastases.
   * AST, ALT <2.5 times the upper limit of normal in patients with evidence of liver metastases.
   * Alkaline phosphatase <2.5 times the upper limit of normal in patients with evidence of hepatic metastases
   * Values of serum creatinine < 1.5 mg / dl. - CCr ( Creatinine Clearance rate) ≥ 60 mL / min 9 . During the study of male and female patients must use adequate contraceptive methods .

Exclusion Criteria:

1. Patients with histological evidence of malignant insulinoma ( pNET )
2. Surgeries performed within 28 days prior to the start of treatment.
3. Evidence of metastasis at the level of the central nervous system or spinal cord compression . Patients should be subjected to a recent study MRI or CT scan at least 28 days from the date of randomization.
4. Clinically significant cardiovascular disease , such as cardiovascular accidents occurred in less than 6 months, unstable angina , congestive heart failure grade greater than or equal to II according to the classification of the New York Heart Association (NYHA) series cardiac arrhythmias that require treatment.
5. Important comorbidities , metabolic disorders , clinical examination or laboratory investigations , which contraindicate the use of drugs to study, or patients at high risk of complications from the treatment.
6. Active or uncontrolled severe infections .
7. Cirrhosis , acute hepatitis or chronic active hepatitis .
8. Poor control of diabetes HbA1c > = 8.0 % .
9. Diabetic patients who are treated with metformin are eligible if they have enabled the treatment with metformin for less than 6 months. Are excluded diabetic patients who make use of other hypoglycemic agents such as sulfonylureas, insulin , glinides as monotherapy or in combination with metformin.
10. Using anti - IL6 (Interleukin 6) or IGF1 .
11. Uncontrolled high blood pressure , atrial fibrillation .
12. History of immunosuppression included positive HIV test .
13. No previous or concomitant oncological pathology , except: basal cell skin cancer, in situ , as long as every other cancer patient diseasefree for at least 5 years.
14. They excluded patients with a condition of metabolic acidosis , acute or chronic , including ketoacidosis .
15. History of alcohol abuse , or habitual intake of alcohol (≥ 3 glasses of alcoholic drinks / day) sufficient to cause hepatotoxicity.
16. Prolonged fasting .
17. Severe states of dehydration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-06; Primary Completion 2021-06 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
to determine the progression free survival rate (PFS) at 12 months from the first drug administration in patients with advanced pancreatic neuroendocrine tumors | 1 year
  progression free survival rate at 12th month of treatment, according to RECIST criteria version 1.0

SECONDARY OUTCOMES:
to determine the safety and tolerability of the combination of Everolimus, Octreotide LAR and Metformin as measured according to the National cancer Institute-Common Toxicity Criteria v. 3.0 guidelines | 1 year
  safety is measured according to the National cancer Institute-Common Toxicity Criteria v. 3.0 guidelines
to determine the overall survival of the combination of Everolimus, Octreotide LAR and Metformin. | 3 years
  overall survival is defined as the time interval between enrollment and the date of the death from any cause.
to determine the response rate of the combination of Everolimus, Octreotide LAR and Metformin. | 1 year
  response rate is defined as the percentage of patients presenting objective responce of the disease, according to RECIST Criteria version 1.0.
to determine the biochemical response of the combination of Everolimus, Octreotide LAR and Metformin. | 1 year
  the biochemical response is defined as the impact of study treatment on general neuroendocrine tumors biomarkers, Chromogranine A and Enolase neuron specific and circulating plasma IL6, IL8 and IGF-1 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Filippo De Braud, MD, Principal Investigator — INT MILANO; Roberto Buzzoni, MD, Principal Investigator — INT MILANO; Sara Pusceddu, MD, Principal Investigator — INT MILANO
Locations (1):
- Fondazione IRCCS Istituto Tumori Milano, Milan, Italy

REFERENCES:
- [Derived] Pusceddu S, de Braud F, Concas L, Bregant C, Leuzzi L, Formisano B, Buzzoni R. Rationale and protocol of the MetNET-1 trial, a prospective, single center, phase II study to evaluate the activity and safety of everolimus in combination with octreotide LAR and metformin in patients with advanced pancreatic neuroendocrine tumors. Tumori. 2014 Nov-Dec;100(6):e286-9. doi: 10.1700/1778.19298. PMID 25688512